CLINICAL TRIAL: NCT01100996
Title: The Effect of Enriched Enteral Nutrition on Inflammation and Sub-clinical Organ Dysfunction During Human Endotoxemia
Brief Title: Anti-inflammatory Effects of Enriched Enteral Nutrition During Human Experimental Endotoxemia
Acronym: VIHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Prof. Dr. J.G. van der Hoeven, Radboud University Nijmegen Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009/168
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2010-02

CONDITIONS: Endotoxemia
Keywords: enteral nutrition; endotoxemia; innate immunity; nutritional anti-inflammatory pathway; intestinal damage
MeSH Terms: conditions — Endotoxemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- fasted control (No Intervention): Volunteers are fasted for 10 hours and subjected to experimental endotoxemia
- control feeding (Placebo Comparator): Volunteers are fed a control nutrition starting 1 hour prior to LPS administration until 6 hours after LPS
  Interventions: Other: control enteral nutrition
- enriched feeding (Active Comparator): volunteers receive the investigational feeding starting 1 hour prior to LPS administration until 6 hours after LPS
  Interventions: Other: enriched enteral feeding

INTERVENTIONS:
Other: control enteral nutrition — This feeding consists of 20en% fat, 16en% protein and 49en% carbohydrates
  Arms: control feeding
Other: enriched enteral feeding — This feeding contains 46 energy percent (en%) fat, 24en% protein and 30en% carbohydrates and is enriched with phospholipids.
  Arms: enriched feeding

SUMMARY:
During sepsis and septic shock the immune response can be overwhelming leading to excessive tissue damage, organ failure and death. Ideally, the inflammatory response is modulated leading to both adequate protection to invading pathogens as well as limitation of an exuberant immune response. In the last years, experimental evidence has been accumulating that enteral administration of lipid-enriched nutrition attenuates inflammation and preserves organ integrity in several inflammatory models. The current study investigates the immune-modulating potential of enriched enteral nutrition in a human setting of experimental endotoxemia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 35 yrs
* Male
* Written informed consent
* non-smoking

Exclusion Criteria:

* Use of any medication (e.g. NSAID's, antibiotics, gastrointestinal motility altering medicine, corticosteroids)
* Smoking in the past year
* History, signs or symptoms of cardiovascular disease
* (Family; first degree) history of cerebrovascular disease
* Previous vagal collapse
* Hypertension (defined as RR systolic > 160 or RR diastolic > 90)
* Hypotension (defined as RR systolic < 100 or RR diastolic < 50)
* Renal impairment (defined as plasma creatinin >120 μmol/l)
* Liver enzyme abnormalities ( ASAT > 60 U/L, ALAT > 75 U/L, Gamma-GT > 60 U/L)
* Positive hepatitis serology
* Positive HIV test
* Allergy to milk and/or soy proteins

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
circulating cytokines | several time points from LPS administration until 24 hours

SECONDARY OUTCOMES:
markers for sub-clinical organ damage (kidney, endothelium, intestine) | several time points from LPS administration until 24 h

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Van der Hoeven, PhD, MD, Principal Investigator — Department of Intensive Care Medicine, Radboud University Nijmegen Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

REFERENCES:
- [Background] Luyer MD, Greve JW, Hadfoune M, Jacobs JA, Dejong CH, Buurman WA. Nutritional stimulation of cholecystokinin receptors inhibits inflammation via the vagus nerve. J Exp Med. 2005 Oct 17;202(8):1023-9. doi: 10.1084/jem.20042397. Epub 2005 Oct 10. PMID 16216887
- [Background] Luyer MD, Derikx JP, Beyaert R, Hadfoune M, van Kuppevelt TH, Dejong CH, Heineman E, Buurman WA, Greve JW. High-fat nutrition reduces hepatic damage following exposure to bacterial DNA and hemorrhagic shock. J Hepatol. 2009 Feb;50(2):342-50. doi: 10.1016/j.jhep.2008.08.025. Epub 2008 Nov 8. PMID 19070388
- [Background] de Haan JJ, Lubbers T, Hadfoune M, Luyer MD, Dejong CH, Buurman WA, Greve JW. Postshock intervention with high-lipid enteral nutrition reduces inflammation and tissue damage. Ann Surg. 2008 Nov;248(5):842-8. doi: 10.1097/SLA.0b013e318188752c. PMID 18948813
- [Background] Lubbers T, Luyer MD, de Haan JJ, Hadfoune M, Buurman WA, Greve JW. Lipid-rich enteral nutrition reduces postoperative ileus in rats via activation of cholecystokinin-receptors. Ann Surg. 2009 Mar;249(3):481-7. doi: 10.1097/SLA.0b013e318194d187. PMID 19247038